CLINICAL TRIAL: NCT01441778
Title: Efficacy of Buffered Hypertonic Saline Nasal Irrigation in Children With Symptomatic Allergic Rhinitis : A Randomized Double-blind Study.
Brief Title: Efficacy of Buffered Hypertonic Saline(BHS)Nasal Irrigation in Allergic Rhinitis (AR) Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, araya satdhabudha, clinical professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-PE-2-CR038-038/53; 14/2553 (Other Grant/Funding Number: Thammasat research grant)
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Rhinitis
Keywords: nasal irrigation; allergic rhinitis; children
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSS irrigation salt (Active Comparator)
  Interventions: Drug: NSS nasal irrigation salt
- BHS nasal irrigaiton salt (Experimental)
  Interventions: Drug: BHS nasal irrigation salt

INTERVENTIONS:
Drug: NSS nasal irrigation salt — nasal irrigation twice daily for 4 weeks period
  Other Names: NORMALINE
  Arms: NSS irrigation salt
Drug: BHS nasal irrigation salt — nasal irrigation twice daily for 4 weeks period
  Other Names: SEANIS
  Arms: BHS nasal irrigaiton salt

SUMMARY:
The purpose of this study is to investigate whether buffered hypertonic saline (BHS) is superior to normal saline (NSS) for improving mucociliary function and relief nasal symptoms in children with allergic rhinitis.

DETAILED DESCRIPTION:
1. BHS is superior to NSS for improving mucociliary function that by measure saccharine clearance time(SCT)at 10 minute after nasal irrigation compare to baseline.
2. BHS is superior to NSS for clinical effectiveness at short period and 1 month follow up

   * at short period: compare the following results at baseline and 10 minute after nasal irrigation

     1. total nasal symptom score(TNSS)
     2. satisfaction to nasal irrigation
     3. side effect
   * at 2 and 4 weeks follow up : compare the following results at baseline and 10 minute after nasal irrigation

     1. quality of life(by specific questionnaire for Thai allergic rhinoconjunctivitis patient)
     2. medication use to relieve AR symptom(from diary record)
     3. compliance for nasal irrigation (from diary record)
     4. side effect (from diary record)
     5. overall satisfaction to nasal irrigation

ELIGIBILITY:
Inclusion Criteria:

1. age 6-15 years
2. diagnosed AR obtained by history, physical examination and positive skin prick test or nasal cytology
3. TNSS ≥ 4 at the first visit of this study

Exclusion Criteria:

1. Patients with a history of nasal anatomical defects
2. Abnormal nasal ciliary function or an upper respiratory tract infection in the preceding 2 weeks

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The change from baseline in SCT at 10 minute after nasal irrigation of BHS and NSS | baseline, 10 minute after nasal irrigaiton
  SCT method : subjects seated with their head upright. A rhinoprobe was used to place a small piece of saccharine on the medial aspect of the inferior turbinate approximately 1 cm, posterior to the nasal vestibule. The SCT was recorded as the subject's first perception of a sweet taste.

SECONDARY OUTCOMES:
The effect of BHS and NSS on clinical effectiveness | 1st visit, 2nd week and 4 week follow up
  evaluate total nasal symptom score, side effect, satisfaction for nasal irrigation, quality of life at 1st visit, 2nd week and 4 week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Araya Satdhabudh, MD, Principal Investigator — Thammasat University
Locations (1):
- Araya Satdabudha, Klong Luang, Pratumthanee, Thailand